CLINICAL TRIAL: NCT06885814
Title: A Phase II Clinical Study on the Efficacy and Safety of Adebrelimab Combined With Chemoradiotherapy in Patients With Unresectable Locally Advanced or Postoperative Recurrent Esophageal Squamous Cell Carcinoma
Brief Title: Efficacy and Safety of Adebrelimab Combined With Chemoradiotherapy in Patients With Unresectable Locally Advanced or Postoperative Recurrent Esophageal Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2024-242
Record Dates: First submitted 2025-03-02; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Unresectable; locally advanced; postoperative recurrent; esophageal squamous cell carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adebrelimab combined with chemoradiotherapy (Experimental)
  Interventions: Drug: Adebrelimab: 20mg/kg day1, Q3W, 3 times

INTERVENTIONS:
Drug: Adebrelimab: 20mg/kg day1, Q3W, 3 times — Concurrent Chemoradiotherapy combined with Immunotherapy，including： Radiotherapy: intensity modulated radiotherapy, PGTV 50-50.4Gy/25-28F, 1.8-2Gy/F, 5 times a week; Chemotherapy: paclitaxel 50mg/ m2 + cisplatin 25mg/ m2, intravenous infusion of day1, once a week, a total of 5 times; Adebrelimab: 20mg/kg day1, Q3W, 3 times.

SUMMARY:
This study was a single-center, single-arm, open-label phase II clinical trial. Thirty patients with unresectable locally advanced or postoperative recurrent esophageal squamous cell carcinoma were treated with concurrent chemoradiotherapy combined with immunotherapy. The radiotherapy regimen was intensity-modulated radiotherapy with PGTV at 50-50.4 Gy/25-28 fractions, 1.8-2 Gy per fraction, five times a week. The chemotherapy regimen was paclitaxel 50 mg/m2 and cisplatin 25 mg/m2 intravenous infusion on day 1, once a week for five times. The immunotherapy was with adebutilimab at 20 mg/kg on day 1, every three weeks for three times. One week before radiotherapy, gastroscopy, chest CT or PET-CT images were taken as the baseline standard. Based on the results of gastroscopy, chest CT or PET-CT before and after treatment, the number of patients with complete response (CR), partial response (PR), stable disease (SD) and progressive disease (PD) in the two groups was observed. The objective response rate (ORR) was calculated as CR + PR, and the disease control rate (DCR) was calculated as CR + PR + SD. The progression-free survival (PFS), overall survival (OS), 1-year and 2-year survival rates and adverse reactions were also statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old, gender unlimited
2. Esophageal squamous cell carcinoma confirmed by histology and unresectable locally advanced or postoperative recurrence
3. According to the solid tumor efficacy evaluation criteria (RECIST1.1), there is at least one measurable lesion; And the lesion had not received prior radiotherapy
4. ECOG: 0~1
5. Expected survival ≥12 weeks 6. Laboratory examination: neutrophils ≥1.5 x 109/L, platelets ≥100 x 109/L; Hemoglobin ≥ 9g/L; Albumin ≥ 2.8g/dL; Bilirubin ≤1.5 times ULN, ALT and AST≤2.5 times ULN

7: Subjects voluntarily joined the study, signed informed consent, had good compliance, and cooperated with follow-up 8: Tissue samples should be provided for biomarker analysis such as (PD-L1). Newly acquired tissues are preferred, and 15 5-6um thick paraffin sections can not be provided for archiving by the recent organizer

Exclusion Criteria:

1. Other malignant tumors have been diagnosed within the previous 5 years
2. There is distant organ metastasis (according to AJCC stage, supraclavicular lymph node metastasis is M1, which should be excluded)
3. Lesions invading the trachea or large blood vessels, or investigators judge that there is a high risk of esophageal/tracheal fistula or bleeding
4. Have any history of active autoimmune disease or autoimmune disease
5. Have clinical symptoms or diseases of the heart that are not under control
6. Active infection or fever (except definite tumor fever)
7. History or evidence of interstitial lung disease or active non-infectious pneumonia
8. Patients with immune dysfunction and active hepatitis
9. Those who have previously received PD-1 or PD-L1 antibody therapy
10. Allergic to any drug in this protocol
11. Patients receiving immunosuppressive drugs or corticosteroids >10mg/ day of prednisone therapeutic dose within 14 days prior to enrollment
12. Patients who had received radiotherapy, chemotherapy, targeted therapy, or immunotherapy within 4 weeks prior to enrollment
13. Pregnant or lactating women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-06 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate at 3 months after radiotherapy (ORR) | Three months after radiation
  ORR includes Complete Response (CR) and Partial Response (PR) according to accepted response evaluation criteria (such as solid tumor RECIST version 1.1), (1) Complete response (CR) : Except for nodular disease, all target lesions disappeared completely. All target nodules must be reduced to normal size (short axis < 10 mm). All target lesions must be evaluated. (2) Partial response (PR) : Total diameter of all measurable target lesions is ≥ 30% below baseline. The short diameter was used for the sum of the target nodules, while the longest diameter was used for the sum of all other target lesions. All target lesions must be evaluated.

SECONDARY OUTCOMES:
Overall survival | From the date of treatment initiation (or diagnosis) to the date of death from any cause, assessed up to 120 months
Progression free survival | The time from the start of treatment to tumor progression or death due to any cause， assessed up to 120 months
Clinical complete response rate | "Monitored throughout the treatment period and during follow-up, an average of 2 years"
  Except for nodular disease, all target lesions disappeared completely. All target nodules must be reduced to normal size (short axis < 10 mm). All target lesions must be evaluated
Quality of life scores of cancer patients | "Monitored throughout the treatment period and during follow-up, an average of 2 years
  Assess the patient's physical function, psychological state, social function, symptom burden, and overall health status through telephone follow-ups, return visits for review, and other methods .The measurement tool is SF-36 Quality of Life Assessment Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No